CLINICAL TRIAL: NCT00831389
Title: Effect of Closed Loop Glucose Control on Exercise-Associated Hypoglycemia
Acronym: ePID-03
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ePID-03
Record Dates: First submitted 2009-01-26; First posted 2009-01-28 (Estimated); Results first posted 2012-10-11 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Closed Loop (CL) Phase (Experimental): Closed Loop (CL) Phase
  Interventions: Device: Closed Loop
- Standard of Care (OL) Phase (No Intervention): Standard of Care (OL) Phase or Open Loop Phase

INTERVENTIONS:
Device: Closed Loop — Insulin pump controlled by closed loop unit and algorithm
  Arms: Closed Loop (CL) Phase

SUMMARY:
The purpose of the study is to compare the glycemic control during and following aerobic exercise using either an open or closed-loop insulin delivery system.

DETAILED DESCRIPTION:
This is an open-label, single-center, randomized crossover study evaluating the performance of a closed-loop insulin delivery system using a subcutaneous glucose sensor and an external insulin pump and comparing it to an open-loop delivery system during aerobic exercise. Subject participation will be for a maximum of 16 weeks including an outpatient study (up to 6 days) and two inpatient studies (one closed-loop; the other open-loop). The closed- and open-loop visit consists of approximately 67 hours over 4 days and 3 nights.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 12-30 years of age.
* Subjects must weigh at least 50 kg to accommodate phlebotomy.
* Previously diagnosed Type 1 Diabetes Mellitus
* Diabetes duration at least 1 year.
* Currently treating their diabetes with an insulin pump.
* A1C of ≤ 9.0 % at time of enrollment.
* Willing to have an intravenous (IV) line inserted for frequent blood sampling and infusion of glucose if needed.
* Willing to wear two (2) subcutaneous glucose sensors and two (2) transmitters simultaneously during closed-loop portion of the study.
* Be in good general health without other acute or chronic illnesses except treated hypothyroidism or celiac disease and asthma not requiring glucocorticoid use.
* Able to tolerate a 75-minute exercise period of moderate intensity.
* Speak and understand English.
* Subject and parent (if minor) must be able to comprehend and sign the informed consent form and other study documents.

Exclusion Criteria:

* Pregnancy (urine pregnancy test) or lactation, if female.
* Subject has any major concomitant disease or any physical or psychological disorder within the last five years, which might be considered life threatening, or which might confound the collection or interpretation of the study data.
* Subject has a cardiac pacemaker or similar device that may be sensitive to radio frequency telemetry.
* Subject using any of the following medications:

  * glucocorticoids
  * cyclosporine
  * L-asparaginase
  * niacin
  * protease inhibitors
  * anti-psychotics
  * GnRH agonists
  * beta-blockers
  * calcium channel blockers
  * immunosuppressants
  * over-the-counter medications that may effect glucose metabolism.
* Subject has any of the following conditions

  * insulin allergy
  * severe insulin resistance
  * exercise-induced asthma
  * musculoskeletal problems that may impact ability to complete exercise protocol
  * substance abuse
  * skin ulcers or poor wound healing
  * bleeding disorders
  * chronic infections
  * eating disorders
  * give a history of or are predisposed to major stress
  * any other major organ system disease.
* Subject has experienced two (2) or more severe hypoglycemic events -seizures/coma requiring assistance in the past six (6) months.
* Subject has any other condition that in the investigator's opinion warrants exclusion from the study or precludes him/her from completing the protocol.
* Subjects using dietary supplements within 14 days of study enrollment
* Subject is currently enrolled in another study.

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2009-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Weinzimer, MD, Principal Investigator — Yale University
Locations (1):
- Yale Pediatrics Diabetes Research, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sherr JL, Cengiz E, Palerm CC, Clark B, Kurtz N, Roy A, Carria L, Cantwell M, Tamborlane WV, Weinzimer SA. Reduced hypoglycemia and increased time in target using closed-loop insulin delivery during nights with or without antecedent afternoon exercise in type 1 diabetes. Diabetes Care. 2013 Oct;36(10):2909-14. doi: 10.2337/dc13-0010. Epub 2013 Jun 11. PMID 23757427

RESULTS

PARTICIPANT FLOW:
Groups:
- First Standard of Care or Open Loop, Then CLosed Loop; First Closed Loop, Then Standard of Care or Open Loop: All participants were treated and observed during in-patient visits twice during the study - two (2) in-patient study phases per subject. Each such in-patient phase was conducted for four (4) days. Insulin delivery during the first in-patient study phase was determined by either Standard of Care (OL), or autonomously by a glycemic control algorithm (CL), depending upon randomization. The exercise challenge was conducted on either the second or third day of this visit, depending upon randomization. Insulin delivery during the second in-patient study phase was the delivery mechanism not used during the 1st in-patient visit. The second in-patient study phase exercise challenge was conducted on the day not chosen for exercise during the first in-patient visit. Intervention was performed only when dictated by protocol or determined necessary by the Health Care Professionals monitoring the study.
Period: Overall Study
Arm/Group | First Standard of Care or Open Loop, Then CLosed Loop | First Closed Loop, Then Standard of Care or Open Loop
Started | 6 | 7
Completed | 6 | 6
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- First Closed Loop, Then Standard of Care or Open Loop: First Closed Loop, Then Standard of Care or Open Loop
- First Standard of Care or Open Loop, Then CLosed Loop: First Standard of Care or Open Loop, Then CLosed Loop
- Total: Total of all reporting groups
Arm/Group | First Closed Loop, Then Standard of Care or Open Loop | First Standard of Care or Open Loop, Then CLosed Loop | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 4 | 11
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.4 (2.1) | 17.7 (4.7) | 15.9 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Plasma Glucose (PG) Response to Exercise
Description: PG at start of exercise minus the subsequent PG nadir
Time Frame: Begins at start of exercise, at or after 15:00 on the in-patient visit day randomly assigned each subject for exercise; ends at start of the subsequent meal. Median period: 121 minutes (min), interquartile range (IQR): 15 min, range: 93 to 133 min.
Population: All subjects were used for final analysis
Measure: Median (Inter-Quartile Range); unit: mg/dL
Groups:
- Standard of Care (OL) Phase: Four day inpatient visit during which insulin administration was dictated by standard of care. Subject determines basal rate, meal bolusing, and any correction boluses using her/his normal regimen. Health Care Provider intervention only when dictated by protocol or determined necessary by the Health Care Professionals monitoring the study.
- Closed Loop (CL) Phase: Four day inpatient visit during which insulin administration was determined autonomously by a glycemic control algorithm, with the exception of pre-meal bolus determined by study protocol. Subject performs no adjustment to insulin dosage. Health Care Provider intervention only when dictated by protocol or determined necessary by the Health Care Professionals monitoring the study.
Arm/Group | Standard of Care (OL) Phase | Closed Loop (CL) Phase
Number analyzed (Participants) | 12 | 12
mg/dL | 75 [48 to 100] | 90.5 [59.75 to 105]
Statistical Analysis 1: Comparison: Standard of Care (OL) Phase vs Closed Loop (CL) Phase; Null hypothesis: Median change in PG concentration due to exercise for the OL and CL study phases do not differ; Test type: Superiority or Other; p = 0.791, Wilcoxon (Mann-Whitney) — p < 0.05 is considered significant

2. Primary Outcome: Incidence of Hypoglycemia Immediately Following Exercise
Description: Tally of episodes where either plasma glucose (PG) < 60 mg/dL, or supplemental glucose was administered to prevent imminent PG < 60 mg/dL. Maximum tally of hypoglycemic events within any 30 minute period is 1.
Time Frame: Begins at end of exercise, at or after 16:15 on the in-patient visit day randomly assigned each subject for exercise; ends at 22:00 of same day. Median period: 333 minutes (min), interquartile range (IQR): 28 min, range: 262 to 344 min.
Population: All subjects were used for final analysis
Measure: Median (Inter-Quartile Range); unit: hypoglycemic events
Arm/Group | Standard of Care (OL) Phase | Closed Loop (CL) Phase
Number analyzed (Participants) | 12 | 12
hypoglycemic events | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Standard of Care (OL) Phase vs Closed Loop (CL) Phase; Null hypothesis: Median tally of hypoglycemic events immediately following exercise for the OL and CL study phases do not differ; Test type: Superiority or Other; p = 0.5, Wilcoxon (Mann-Whitney) — p < 0.05 is considered significant

3. Primary Outcome: Incidence of Nocturnal Hypoglycemia Following Exercise
Description: as for outcome 2
Time Frame: Begins at 22:00 on the in-patient visit day randomly assigned each subject for exercise; ends at 6:00 of the subsequent day. Period was 480 minutes (min) for all subjects, both study phases.
Population: All subjects were used for final analysis
Measure: Median (Inter-Quartile Range); unit: hypoglycemic events
Arm/Group | Standard of Care (OL) Phase | Closed Loop (CL) Phase
Number analyzed (Participants) | 12 | 12
hypoglycemic events | 0 [0 to 1] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Standard of Care (OL) Phase vs Closed Loop (CL) Phase; Null hypothesis: Median tally of nocturnal hypoglycemic events following exercise for the OL and CL study phases do not differ; Test type: Superiority or Other; p = 0.25, Wilcoxon (Mann-Whitney) — p < 0.05 is considered significant

4. Secondary Outcome: Peak Post-prandial Plasma Glucose (PG)
Description: For each subject and study phase, the six peak PG following each of the six meals were determined. The median of these six peaks became the one peak post-prandial PG value representing each subject and study phase.
Time Frame: Union of 6 meal periods (3 per day on study days 2 & 3). A meal period runs from meal start to start of next meal, or 22:00 for 3rd meal of the day. Union of 6 periods median: 1666 minutes (min), interquartile range (IQR): 15 min, range: 1638 to 1680 min.
Population: All subjects were used for final analysis
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Standard of Care (OL) Phase | Closed Loop (CL) Phase
Number analyzed (Participants) | 12 | 12
mg/dL | 188 [162.5 to 227.875] | 229.75 [207.875 to 242.375]
Statistical Analysis 1: Comparison: Standard of Care (OL) Phase vs Closed Loop (CL) Phase; Null hypothesis: Median peak post-prandial PG for the OL and CL study phases do not differ; Test type: Superiority or Other; p = 0.0669, Wilcoxon (Mann-Whitney) — p < 0.05 is considered significant

5. Secondary Outcome: Nadir Plasma Glucose (PG) Immediately Following Exercise
Description: The PG nadir observed following the start of exercise
Time Frame: as for outcome 1
Population: All subjects were used for final analysis
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Standard of Care (OL) Phase | Closed Loop (CL) Phase
Number analyzed (Participants) | 12 | 12
mg/dL | 80.5 [65.75 to 120.75] | 70.5 [66.75 to 80.5]
Statistical Analysis 1: Comparison: Standard of Care (OL) Phase vs Closed Loop (CL) Phase; Null hypothesis: Median nadir PG immediately following exercise for the OL and CL study phases do not differ; Test type: Superiority or Other; p = 0.2256, Wilcoxon (Mann-Whitney) — p < 0.05 is considered significant

6. Secondary Outcome: Overnight Nadir Plasma Glucose (PG)
Description: For each subject and study phase, the overnight nadir PG for each of two nights were determined. The mean of these two nadirs became the one nadir overnight PG value representing each subject and study phase.
Time Frame: Union of the two 8-hour overnight periods beginning at 22:00 on in-patient visit days 2 & 3, ending at 6:00 on the subsequent day. The union of the two periods was 960 minutes (min) for all subjects, both study phases.
Population: All subjects were used for final analysis
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Standard of Care (OL) Phase | Closed Loop (CL) Phase
Number analyzed (Participants) | 12 | 12
mg/dL | 74.5 [61.375 to 109.625] | 93.5 [84.5 to 97.25]
Statistical Analysis 1: Comparison: Standard of Care (OL) Phase vs Closed Loop (CL) Phase; Null hypothesis: Median overnight nadir PG for the OL and CL arms do not differ; Test type: Superiority or Other; p = 0.791, Wilcoxon (Mann-Whitney) — p < 0.05 is considered significant

7. Secondary Outcome: Percentage of Time Plasma Glucose (PG) is Within the Euglycemic Range.
Description: For each subject and arm, the percentage of the PG curve such that 70 <= PG curve <= 180 mg/dL. Linear interpolations furnished the data between the actual sampled PG to address potential sample influence bias arising from non-uniform sampling intervals.
Time Frame: Begins at 6:00 of in-patient visit day 2 and ends at 6:00 of day 4; 48 hours total.
Population: All subjects were used for final analysis
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Standard of Care (OL) Phase | Closed Loop (CL) Phase
Number analyzed (Participants) | 12 | 12
percentage of time | 74.1 [66.2 to 81.4] | 79.8 [73.3 to 83.8]
Statistical Analysis 1: Comparison: Standard of Care (OL) Phase vs Closed Loop (CL) Phase; Null hypothesis: Median percentage of time PG is within euglycemic range for the OL and CL phases do not differ; Test type: Superiority or Other; p = 0.2036, Wilcoxon (Mann-Whitney) — p < 0.05 is considered significant

8. Secondary Outcome: Percentage of Time Plasma Glucose (PG) is Above the Euglycemic Range.
Description: For each subject and study phase, the percentage of the PG curve > 180 mg/dL. Linear interpolations furnished the data between the actual sampled PG to address potential sample influence bias arising from non-uniform sampling intervals.
Time Frame: Begins at 6:00 of in-patient visit day 2 and ends at 6:00 of day 4; 48 hours total.
Population: All subjects were used for final analysis
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Standard of Care (OL) Phase | Closed Loop (CL) Phase
Number analyzed (Participants) | 12 | 12
percentage of time | 19.7 [6.7 to 32.6] | 17.3 [15.6 to 21.8]
Statistical Analysis 1: Comparison: Standard of Care (OL) Phase vs Closed Loop (CL) Phase; Null hypothesis: Median percentage of time PG is above euglycemic range for the OL and CL phases do not differ; Test type: Superiority or Other; p = 0.6221, Wilcoxon (Mann-Whitney) — p < 0.05 is considered significant

9. Secondary Outcome: Percentage of Time Plasma Glucose (PG) is Below the Euglycemic Range.
Description: For each subject and study phase, the percentage of the PG curve < 70 mg/dL. Linear interpolations furnished the data between the actual sampled PG to address potential sample influence bias arising from non-uniform sampling intervals.
Time Frame: Begins at 6:00 of in-patient visit day 2 and ends at 6:00 of day 4; 48 hours total.
Population: All subjects were used for final analysis
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Standard of Care (OL) Phase | Closed Loop (CL) Phase
Number analyzed (Participants) | 12 | 12
percentage of time | 6 [0.1 to 10] | 1.1 [0.5 to 2.9]
Statistical Analysis 1: Comparison: Standard of Care (OL) Phase vs Closed Loop (CL) Phase; Null hypothesis: Median percentage of time PG is below euglycemic range for the OL and CL phases do not differ; Test type: Superiority or Other; p = 0.021, Wilcoxon (Mann-Whitney) — p < 0.05 is considered significant

10. Post Hoc Outcome: Overall Incidence of Hypoglycemia
Description: as for outcome 2
Time Frame: Begins at 6:00 of in-patient visit day 2 and ends at 6:00 of day 4; 48 hours total.
Population: All subjects were used for final analysis
Measure: Median (Inter-Quartile Range); unit: hypoglycemic events
Arm/Group | Standard of Care (OL) Phase | Closed Loop (CL) Phase
Number analyzed (Participants) | 12 | 12
hypoglycemic events | 3 [0 to 5.5] | 1 [0.75 to 1]
Statistical Analysis 1: Comparison: Standard of Care (OL) Phase vs Closed Loop (CL) Phase; Null hypothesis: Median tally of hypoglycemic events over 48 hour in-patient period for the OL and CL phases do not differ; Test type: Superiority or Other; p = 0.0176, Wilcoxon (Mann-Whitney) — p < 0.05 is considered significant

ADVERSE EVENTS:
Arm/Group | Standard of Care (OL) Phase | Closed Loop (CL) Phase
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (OL) Phase (N=13) | Closed Loop (CL) Phase (N=13)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less